CLINICAL TRIAL: NCT07020832
Title: A Phase 3, Randomized, Placebo-Controlled, Double-Blinded, Multicenter Study to Evaluate the Efficacy and Safety of Pegcetacoplan in Adults at High Risk of Delayed Graft Function (DGF) Following Kidney Allograft Transplantation
Brief Title: A Phase 3 Study to Evaluate the Efficacy and Safety of Pegcetacoplan in Adults at High Risk of Delayed Graft Function (DGF) Following Kidney Allograft Transplantation
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Apellis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: APL2-DGF-318
Record Dates: First submitted 2025-06-06; First posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Delayed Graft Function; End Stage Renal Disease; Deceased Donor Kidney Transplant
MeSH Terms: conditions — Delayed Graft Function; Kidney Failure, Chronic | interventions — pegcetacoplan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Pegceptacoplan (Active Comparator): Administration as a 20mL IV infusion initially, then as a subcutaneous infusion
  Interventions: Drug: Pegcetacoplan
- Placebo (Placebo Comparator): Administration as a 20mL IV infusion initially, then as a subcutaneous infusion
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Pegcetacoplan — Complement (C3) Inhibitor
  Arms: Pegceptacoplan
Other: Placebo — Sterile solution of equal volume to active arm
  Arms: Placebo

SUMMARY:
A PHASE 3 STUDY TO EVALUATE THE EFFICACY AND SAFETY OF PEGCETACOPLAN IN ADULTS AT HIGH RISK OF DELAYED GRAFT FUNCTION (DGF) FOLLOWING KIDNEY ALLOGRAFT TRANSPLANTATION

ELIGIBILITY:
Inclusion Criteria:

1. Aged at least 18 years
2. Have end-stage kidney disease and be on the waiting list for a kidney transplant from a deceased donor.
3. Be on dialysis at the time of your transplant and produce very little urine (less than 200 mL per day). You must have been on dialysis for at least 3 months.
4. Be receiving your first or second kidney transplant from a deceased donor. If this is your second transplant:

   1. It cannot be due to a serious infection or a serious blood clot in your previous transplant.
   2. Your calculated Panel Reactive Antibody (CPRA) level must be below 50%.
5. Be getting a donor kidney that meets the study's specific requirements.
6. Be at low to medium risk of transplant rejection, and be scheduled to receive:

   1. A medication called ATG as part of your transplant procedure.
   2. Steroids (corticosteroids) as part of your treatment at the time of screening.
   3. A medication called tacrolimus (or a similar drug) after your transplant, according to usual medical practice.
7. Have received certain vaccines before starting the study treatment, specifically:

   1. Pneumococcal (S. pneumoniae)
   2. Meningococcal (N. meningitidis types A, C, W, Y, and B)
   3. Haemophilus influenzae type B

If you haven't had these vaccines, you may still qualify if you're medically shown not to respond to them and your doctor has a plan to give you preventive antibiotics, with the sponsor's approval.

Exclusion Criteria:

1. Have taken part in another medical research study or used an experimental drug, treatment, or device in the past 30 days (or longer, depending on the drug).
2. Have recently used certain medications that affect the immune system, such as rituximab, belimumab, or other approved complement-blocking drugs.
3. Weigh less than 20kg or more than 120kg at screening.
4. Have or had recently had any of the following infections:

   1. Hepatitis B or Hepatitis C (unless treated and no longer active).
   2. HIV (human immunodeficiency virus) at any time.
5. Have had cancer in the past 5 years, unless it was:

   1. A small, treated skin cancer (like basal or squamous cell), or
   2. A very small kidney cancer that was found early and treated.
6. Have received any other organ transplant (except for one previous kidney transplant), or are scheduled for a transplant involving more than one organ.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Time to freedom from dialysis through Day 90 | Duration of dialysis through day 90
  To assess the efficacy of pegcetacoplan compared with that of placebo in participants at high risk of DGF following donor kidney allograft transplant surgery

SECONDARY OUTCOMES:
eGFR at Week 52 | 52 weeks following surgery
  To evaluate the efficacy of pegcetacoplan in reducing the severity of DGF and consequent improvements in short-, medium- and long-term kidney function and kidney allograph outcomes
Proportion of participants with DGF (defined as the need for dialysis in the 7 days posttransplant) | 7 days following surgery
  To evaluate the efficacy of pegcetacoplan in reducing the severity of DGF and consequent improvements in short-, medium- and long-term kidney function and kidney allograph outcomes
eGFR at Day 90 | 90 days following surgery
  To evaluate the efficacy of pegcetacoplan in reducing the severity of DGF and consequent improvements in short-, medium- and long-term kidney function and kidney allograph outcomes
Time to achievement of ≥1200 mL of urine output in a 24-hour period through Day 14 | 14 days following surgery
  To evaluate the efficacy of pegcetacoplan in reducing the severity of DGF and consequent improvements in short-, medium- and long-term kidney function and kidney allograph outcomes
Biopsy-proven rejection-free kidney allograft survival by Week 52 | 52 weeks following surgery
  To evaluate the efficacy of pegcetacoplan in reducing the severity of DGF and consequent improvements in short-, medium- and long-term kidney function and kidney allograph outcomes

IPD SHARING:
Plan to Share IPD: No